CLINICAL TRIAL: NCT07310537
Title: Feasibility of Circulating Tumour DNA (ctDNA) Analysis Using Automated Capillary Blood Sampling
Acronym: ctDNA TAP
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Mirthe Ubink, MD, Erasmus Medical Center
Other Study IDs: NL88018.078.24
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer (Diagnosis); Colorectal Liver Metastasis (CRLM); Circulating Tumor DNA (ctDNA)
Keywords: Colorectal Cancer; Colorectal Liver Metastasis (CRLM); Circulating Tumor DNA (ctDNA); Automated Capillary Blood Sampling
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL venous blood samples will be collected in EDTA tubes, and capillary blood samples will be collected using a K2EDTA Microtainer®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ctDNA TAP: Study Group
  Interventions: Other: Blood Collection - TAP® Device; Other: Blood Collection - Venous

INTERVENTIONS:
Other: Blood Collection - TAP® Device — K2EDTA BD Microtainer
Other: Blood Collection - Venous — 10 mL EDTA Collection Tube

SUMMARY:
The goal of this observational study is to investigate whether circulating tumor-derived DNA (ctDNA) can be reliably detected and analyzed in blood obtained through automated capillary sampling in adult patients (≥21 years) with colorectal liver metastases (CRLM).

The main question it aims to answer is:

* Can ctDNA be detected in small volumes of capillary blood collected using an automated sampling device?
* Do ctDNA levels measured in capillary blood agree with those measured in venous blood from the same patients?

Researchers will compare ctDNA measurements from capillary blood to those from venous blood (reference standard) to see if capillary sampling provides reliable results for ctDNA analysis.

Participants will:

* Provide a small blood sample through automated capillary collection.
* Provide a venous blood sample during the same study visit for comparison.

DETAILED DESCRIPTION:
Rationale: Aging of the general population results in an increasing number of patients who need to be cared for by a decreasing number of health care professionals. To ensure sustainable and patient-centred health care in the near future, rebalanced hospital-based and home-based care is needed. Following surgery of a primary tumour or metastases thereof, patients are offered blood-based follow-up in the hospital, which is necessary to detect recurrence but represents a major burden on the current health care system. The more recently discovered, highly specific circulating tumour-derived DNA fragments (ctDNA) have high potential as a new biomarker and clinical implementation of ctDNA in CRC patient care is expected in the future. However, feasibility of ctDNA detection in blood collected through automated capillary sampling had not yet been investigated.

Objective: to determine the feasibility of ctDNA analysis of blood obtained using automated capillary sampling.

Study design: This proof-of-concept study aims to determine technical feasibility of ctDNA detection in small volumes of capillary blood in 35 patients. Venous blood from the same patients will be used as reference

Study population: All study subjects need to be 21 years or older and provide informed consent to participate in the study. Patients with growing colorectal liver metastases (CRLM) can be included.

Main study endpoint: The primary outcome measure of the study is the agreement between ctDNA measurements in venous versus capillary blood to determine the feasibility of ctDNA analysis through automated capillary blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* A history of histologically confirmed (metastatic) colorectal adenocarcinoma
* Currently diagnosed with (progressive) colorectal liver metastases (CRLM)
* Signed informed consent

Exclusion Criteria:

* Patients who are treated and having a response on chemotherapy, as this may have an effect on the investigated biomarker load
* Illiteracy and/or insufficient proficiency of the Dutch language
* Known medical history of superficial or deep skin infection after venipuncture or intravenous line that required antibiotic treatment and or hospital admittance
* Known medical history of immunodeficiency or current use of medical immunosuppressants
* Known medical history of blood-borne diseases such as, but not limited to, the human immunodeficiency virus, hepatitis and viral hemorrhagic fever

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All study subjects need to be 21 years or older and provide informed consent to participate in the study. Patients with newly diagnosed/and or progressive colorectal liver metastases (CRLM) can be included.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of ctDNA detection in small volumes of capillary blood | Baseline
  This will be investigated through determining the agreement between ctDNA measurements in venous (standard blood collection) versus capillary blood through automated capillary blood sampling. A Kappa >0.75 will be considered as sufficient agreement.

SECONDARY OUTCOMES:
Correlation between ctDNA levels (VAF) in venous and capillary blood | Baseline
  A correlation coefficient of >0.5 will be considered as sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis Verhoef, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC University Medical Center, Rotterdam, South Holland, Netherlands

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT07310537/Prot_SAP_000.pdf